CLINICAL TRIAL: NCT02359539
Title: Marginal Periosteal Pedicle Flap and Platelet Rich Fibrin Barriers for the Treatment of Periodontal Intrabony Defects -Randomized Clinical Trial
Brief Title: Marginal Periosteal Pedicle Flap - Platelet Rich Fibrin Barriers in Treating Periodontal Intrabony Defects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Ahmed Y Gamal, Professor of Periodontology Ain Shams University, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Ain Shams University
Record Dates: First submitted 2014-11-16; First posted 2015-02-10 (Estimated); Last update posted 2015-02-10 (Estimated); Status verified 2014-11

CONDITIONS: Periodontal Pocket
MeSH Terms: conditions — Periodontal Pocket | interventions — Guided Tissue Regeneration

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PRF (Experimental): Platelets rich fibrin,
  Interventions: Procedure: Regenerative therapy
- MPP (Experimental): Marginal periosteal pedicle
  Interventions: Procedure: Regenerative therapy

INTERVENTIONS:
Procedure: Regenerative therapy — Periosteal pedicle, Platelets rich fibrin
  Other Names: Guided tissue regeneration

SUMMARY:
The use of autogenous graft materials has been recorded to be a gold standard in regenerative therapy. This study directed toward evaluation of two autogenous regenerative materials, marginal periosteal pedicle graft (MPP) and platelet rich fibrin (PRF) as membrane barriers for treating intrabony defects. In spite of its reported significant clinical outcomes, the limited availability of the periosteum makes it necessary to evaluate other autogenous alternatives such as PRF that could offer predictable outcomes.

DETAILED DESCRIPTION:
Material and methods: 10 patients with sever chronic periodontitis and at least single ≥4 mm intrabony defect had participated in this randomized clinical study. Subjects were randomly divided into2 groups, Group 1(MPP) defect coverage with xenograft defect fill(10 patients),Group 2(PRF) defect coverage with xenograft defect fill(10 patients).Clinical and radiographic measurements were carried out at 3,6 and 9 months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* No systemic diseases that could influence the outcome of therapy
* Good compliance for plaque control instructions after initial therapy
* Vital teeth
* Had contralateral matched pair of 2- or 3-walled intrabony interproximal defects in premolar or molar teeth
* Probing pocket depth (PPD)≥6 mm and clinical attachment level (CAL) ≥4mm 6) selected 2- or 3-wall intrabony defect depth ≥ 3 mm as detected in diagnostic periapical radiographs,

Exclusion Criteria:

* Pregnant females and patients presented with opened interproximal contact

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2009-08; Primary Completion 2012-04 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Intrabony defect | 9 month after surgery
  measurements of intrabony gain from CEJ to base of defect